CLINICAL TRIAL: NCT06672900
Title: A Multi-Part Phase 1 Study in Healthy Volunteers to Evaluate the Drug-Drug Interaction Potential of Multiple Doses of ALG-000184.
Brief Title: A Multi-part Study of ALG-000184 to Evaluate Safety, Tolerability, Pharmacokinetics and Drug-drug Interaction Potential After Single and Multiple Doses in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALG-000184-204
Record Dates: First submitted 2024-09-25; First posted 2024-11-04 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ALG-000184
MeSH Terms: interventions — Carbamazepine; Itraconazole

STUDY DESIGN:
Intervention Model Description: Open-label, fixed sequence, crossover study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ALG-000184 (Experimental): Single or multiple doses of ALG-000184, an investigational HBV capsid assembly modulator
  Interventions: Drug: ALG-000184
- Carbamazepine (Experimental): Multiple doses of carbamazepine, a strong CYP3A4 inducer, to evaluate potential drug-drug interactions with ALG-000184
  Interventions: Drug: Carbamazepine; Drug: ALG-000184
- Itraconazole (Experimental): Multiple doses of itraconazole, a strong CYP3A4 inhibitor, to evaluate potential drug-drug interactions with ALG-000184.
  Interventions: Drug: Itraconazole (Sporanox); Drug: ALG-000184

INTERVENTIONS:
Drug: Carbamazepine — Commercially available supply.
  Arms: Carbamazepine
Drug: Itraconazole (Sporanox) — Commercially available supply.
  Arms: Itraconazole
Drug: ALG-000184 — Study Investigational Product

SUMMARY:
This Phase 1 study consists of two parts, all conducted in healthy volunteers (HVs).

In Part 1, the drug-drug interaction (DDI) potential of ALG-000184 will be explored with Itraconazole; participants will be assigned to receive multiple doses of ALG-000184 and Itraconazole over a two week period.

In Part 2, the drug-drug interaction (DDI) potential of ALG-000184 will be explored with Carbamazepine; participants will be assigned to receive multiple doses of ALG-000184 and ascending doses of Carbamazepine over an 18 day period.

The 2 parts may be conducted in parallel.

ELIGIBILITY:
Inclusion Criteria for All Participants:

1. Male or female between 18 and 55 years of age.
2. BMI 18.0 to 32.0 kg/m^2
3. Female participants must have a negative serum pregnancy test at screening.
4. Subjects must have a 12-lead electrocardiogram (ECG) that meets the protocol criteria.

Exclusion Criteria for All Participants:

1. Participants with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation.
2. Participants with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Participants with a history of clinically significant drug allergy.
4. Participants with excessive use of alcohol defined as regular consumption of ≥14 standard drinks/week (US CDC 2022)
5. Participants that are unwilling to abstain from alcohol use for 1 week prior to start of the study through end of study follow up.
6. Participants with positive results for urine drug screen, alcohol or cotinine test at screening and Day -1.
7. Participants with Hepatitis A, B, C, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection.
8. Participants with sensitivity to CYP3A4 or P-gp substrates, inhibitors/inducers.
9. Participants with clinically significant abnormal vital signs or physical examination.
10. Participants with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m^2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-07-07 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of itraconazole (Part 1)
Area under the concentration time curve [AUC] | Up to 29 days.
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)
Time to maximum plasma concentration [Tmax] | Up to 29 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)
Time to maximum plasma concentration [Tmax] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Itraconazole (Part 1)
Maximum plasma concentration [Cmax] | Up to 29 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)
Maximum plasma concentration [Cmax] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Itraconazole (Part 1)
Minimum plasma concentration [Cmin] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of itraconazole (Part 1)
Minimum plasma concentration [Cmin] | Up to 29 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)
C0 [predose] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of itraconazole (Part 1)
C0 [predose] | Up to 29 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)
Half-life [t1/2] | Up to 24 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of itraconazole (Part 1)
Half-life [t1/2] | Up to 29 days
  Pharmacokinetic parameters of ALG-001075 and metabolite ALG-000302 after multiple doses of Carbamazepine (Part 2)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 days for Part 1
  The number and severity of treatment emergent adverse events in up to n=24 participants as assessed by DAIDS v2.1(July 2017)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 29 days for Part 2
  The number and severity of treatment emergent adverse events in up to n=24 participants as assessed by DAIDS v2.1(July 2017)
Mean Change from Baseline QTc at different exposure levels | Up to 24 days for Part 1.
  Evaluate the concentration-QT relationship of ALG-000175 and metabolite ALG-000302 to determine the QTc prolongation potential of ALG-000184.
Mean Change from Baseline QTc at different exposure levels | Up to 29 days for Part 2.
  Evaluate the concentration-QT relationship of ALG-000175 and metabolite ALG-000302 to determine the QTc prolongation potential of ALG-000184.

OTHER OUTCOMES:
Cholesterol | Up to 24 days in Part 1
  Intends to monitor plasma samples from baseline to measure 4-β-hydroxycholesterol, an induction marker of CYP450.
Cholesterol | Up to 29 days in Part 2
  Intends to monitor plasma samples from baseline to measure 4-β-hydroxycholesterol, an induction marker of CYP450.
Area under the concentration time curve [AUC] | 29 days
  Pharmacokinetic parameters of Carbamazepine and applicable metabolite
Area under the concentration time curve [AUC] | 24 days
  Pharmacokinetic parameters of itraconazole and applicable metabolite
Maximum plasma concentration [Cmax] | 24 days
  Pharmacokinetic parameters of Itraconazole and applicable metabolite
Maximum plasma concentration [Cmax] | 29 days
  Pharmacokinetic parameters of Carbamazepine and applicable metabolite
Minimum plasma concentration [Cmin] | 24 days
  Pharmacokinetic parameters of Itraconazole and applicable metabolite
Minimum plasma concentration [Cmin] | 29 days
  Pharmacokinetic parameters of Carbamazepine and applicable metabolite
C0 [predose] | 24 days
  Pharmacokinetic parameters of Itraconazole and applicable metabolite
C0 [predose] | 29 days
  Pharmacokinetic parameters of Carbamazepine and applicable metabolite
Half-life [t1/2] | 24 days
  Pharmacokinetic parameters of Itraconazole and applicable metabolite
Half-life [t1/2] | 29 days
  Pharmacokinetic parameters of Carbamazepine and applicable metabolite
Time to maximum plasma concentration [Tmax] | 24 Days
  Pharmacokinetic parameters of Itraconazole and applicable metabolite
Time to maximum plasma concentration [Tmax] | 29 days
  Pharmacokinetic parameters of carbamazepine and applicable metabolite

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided